CLINICAL TRIAL: NCT00681889
Title: Effectiveness and Safety of Topical Ranibizumab for Treatment of Corneal Neovascularization (NV)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reza Dana, MD (Other)
Responsible Party: Sponsor-Investigator, Reza Dana, MD, Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-11-069; 07-11-069 (Other: Massachusetts Eye and Ear Infirmary)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-10

CONDITIONS: Corneal Neovascularization
MeSH Terms: conditions — Corneal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): 10 Patients will receive treatment (Ranibizumab)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 10 Patients will receive treatment (Ranibizumab)
  Other Names: Lucentis

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of ranibizumab (Lucentis) in treatment of corneal neovascularization.

DETAILED DESCRIPTION:
This is an open label, single site, uncontrolled, single group assignment, safety/efficacy, Phase I study of topical administered ranibizumab in subjects with corneal neovascularization. Ten eyes of patients with corneal neovascularization will be recruited. Patients with superficial or deep corneal neovascularization that extends farther than 2 mm from the limbus will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years old
* Patients with superficial or deep corneal neovascularization that extends farther than 2 mm from the limbus

Exclusion Criteria:

* Has received investigational therapy within 60 days prior to study entry
* Has received treatment with anti-VEGF agents (intraocular or systemic) within 45 days of study entry
* Concurrent use of systemic anti-VEGF agents
* Full thickness or lamellar keratoplasty within 90 days prior to study entry
* Ocular surface reconstruction within 90 days prior to study entry
* Other ocular surgeries within 90 days prior to study entry
* Corneal or ocular surface infection within 90 days prior to study entry
* Ocular or periocular malignancy
* Contact lens (excluding bandage contact lens) within 30 days prior to study entry
* Persistent epithelial defect (>1mm2 and ≥14 days duration) within 30 days prior to study entry
* Systemic, intravitreal, or periocular steroids within 30 days prior to study entry
* Change in dose/frequency of topical steroids and/or NSAIDs within 30 days prior to study entry
* Hypertension: systolic BP > 150 or diastolic BP > 90
* History of thromboembolic event within 6 months prior to study entry
* Current diagnosis of diabetes, Pregnancy (positive pregnancy test) or lactation
* Premenopausal women not using adequate contraception (The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch)
* Participation in another simultaneous medical investigation or trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Dana, M.D., MPH, Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Cornea Service at the Massachusetts Eye and Ear Infirmary from April 2008 through September 2009.
Pre-assignment Details: Participants were assigned to the investigational treatment upon a full eligibility screening. Participants were not eligible if they had received investigational therapy within 60 days, received treatment with anti-VEGF agents (intraocular or systemic) within 45 days, were concurrently using systemic anti-VEGF agents amongst other criteria.
Groups:
- Treatment Arm: 10 eyes of 9 patients will receive treatment (Ranibizumab)
  Ranibizumab : 10 eyes of 9 patients will receive treatment (Ranibizumab)
Period: Overall Study
Arm/Group | Treatment Arm
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: 10 Patients will receive treatment (Ranibizumab)
  Ranibizumab : 10 Patients will receive treatment (Ranibizumab)
Arm/Group | Treatment Arm
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular Adverse Event
Description: Incidence and severity of ocular adverse events, as identified by eye examination and visual acuity testing
Time Frame: 16 Weeks
Population: All participants enrolled into the study were analyzed.
Measure: Number; unit: participants
Groups:
- Treatment Arm: 9 Patients will receive treatment (Ranibizumab)
  Ranibizumab : 9 Patients will receive treatment (Ranibizumab)
Arm/Group | Treatment Arm
Number analyzed (Participants) | 9
participants | 0

2. Primary Outcome: Incidence and Severity of Other Adverse Events, as Identified by Physical Examination, Subject Reporting, and Changes in Vital Signs
Time Frame: 16 Weeks
Reporting Status: Not Posted

3. Secondary Outcome: Efficacy by Comparison Size and Extent of Blood Vessels in Baseline and Follow-up Corneal Photographs
Time Frame: Prospective
Reporting Status: Not Posted

4. Secondary Outcome: Efficacy by Measuring Mean Change of BCVA
Time Frame: Prospective
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
Further and larger studies are needed to better establish the efficacy profile of this drug and optimize its dosing and formulation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes